CLINICAL TRIAL: NCT06931340
Title: Docetaxel Addition in Metastatic Castrate-Sensitive Prostate Cancer (ASPIRE)
Brief Title: Testing the Addition of Docetaxel (Chemotherapy) to the Usual Treatment (Hormonal Therapy and Apalutamide) for Metastatic Prostate Cancer, ASPIRE Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A032302; NCI-2025-00838 (Other: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Castration-Sensitive Prostate Carcinoma; Metastatic Prostate Adenocarcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Docetaxel; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (ADT, apalutamide) (Active Comparator): Patients receive ADT at the discretion of the investigator and apalutamide PO QD. Cycles repeat every 12 weeks in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT scan or MRI and bone scan throughout the study. Patients may optionally undergo PSMA-PET scans and blood sample collection throughout the study.
  Interventions: Drug: Androgen Therapy; Drug: Apalutamide; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Bone Scan; Procedure: PSMA PET Scan; Procedure: Biospecimen Collection; Other: Questionnaire Administration
- Arm 2 (ADT, apalutamide, docetaxel) (Experimental): Patients receive ADT at the discretion of the investigator and apalutamide PO QD. Cycles repeat every 12 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive docetaxel IV over 1 hour every 21 days for up to 6 doses. Additionally, patients undergo CT scan or MRI and bone scan throughout the study. Patients may optionally undergo PSMA-PET scans and blood sample collection throughout the study.
  Interventions: Drug: Androgen Therapy; Drug: Apalutamide; Drug: Docetaxel; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Bone Scan; Procedure: PSMA PET Scan; Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Androgen Therapy — Given ADT
Drug: Apalutamide — Given PO
Drug: Docetaxel — Given IV
  Other Names: Taxotere
  Arms: Arm 2 (ADT, apalutamide, docetaxel)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT Scan; CT Scan
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI
Procedure: Bone Scan — Undergo Bone Scan
Procedure: PSMA PET Scan — Undergo PSMA PET Scan
Procedure: Biospecimen Collection — Undergo blood sample collection
Other: Questionnaire Administration — undergo Questionnaire Administration

SUMMARY:
This phase III trial compares the effect of adding docetaxel to hormonal therapy and apalutamide versus hormonal therapy and apalutamide alone in treating patients with prostate cancer that has spread from where it first started (primary site) to other places in the body (metastatic). Docetaxel is in a class of medications called taxanes. It stops tumor cells from growing and dividing and may kill them. Hormone therapy for prostate cancer, also called androgen deprivation therapy (ADT), uses surgery or drugs to lower the levels of male sex hormones in a man's body. This helps slow the growth of prostate cancer. Apalutamide is in a class of medications called androgen receptor inhibitors. It works by blocking the effects of androgen (a male reproductive hormone) to stop the growth and spread of tumor cells. Giving docetaxel in addition to the usual treatment of hormonal therapy and apalutamide may work better in treating patients with metastatic prostate cancer than the usual treatment alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the addition of docetaxel to androgen deprivation therapy and apalutamide improves overall survival for men with metastatic castrate sensitive prostate cancer.

SECONDARY OBJECTIVES:

I. To determine if the addition of docetaxel to androgen deprivation therapy and apalutamide improves overall survival for men whose cancers have loss or inactivating mutations of TP53, PTEN, or RB1.

II. To determine if the addition of docetaxel to ADT plus apalutamide improves the time to radiographic progression per Prostate Cancer Working Group 3 (PCWG3) guidelines.

III. To determine the time to castration-resistant prostate cancer (CRPC) between arms.

IV. To determine symptomatic skeletal event free survival (SSE-FS) between arms.

V. To determine the safety and tolerability of the triplet versus doublet using Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.

VI. To determine radiographic progression free survival (rPFS), and overall survival (OS) in patients by the stratification factors a) volume/timing of disease (metachronous high volume, synchronous high volume, and synchronous low volume metastases on conventional imaging) and b) tumor suppressor gene alteration status (0 versus [vs] 1 vs 2+) between arms.

VII. To determine prostate specific antigen (PSA) 90 response rate at 6 weeks and 6 months between arms.

VIII. To determine time to PSA progression by PCWG3 criteria between arms. IX. To determine objective response rate (ORR) in patients with measurable disease between arms.

EXPLORATORY OBJECTIVES:

I. To determine the time to worsening of physical symptoms of disease based on functional assessment of cancer therapy/National Comprehensive Cancer Network prostate cancer symptom index 17 item questionnaire (NCCN-FACT FPSI-17) between arms.

II. To compare quality of life as measured by Functional Assessment of Cancer Therapy-Prostate (FACT-P) trial outcome index in patients with metastatic castrate-sensitive prostate cancer (mCSPC) who receive ADT + apalutamide + docetaxel vs ADT + apalutamide at the 24-month time point.

III. To compare quality of life as measured by other scales of the FACT-P in the two arms.

IV. To compare quality of life as measured by FACT-P total outcome index in the two arms at other timepoints.

V. To compare pain severity and interference as measured by the Brief Pain Inventory Short Form (BPI-SF) in the two arms.

VI. To compare quality-adjusted life years which accounts for survival and utility (measured by European Quality of Life Five Dimension Five Level Scale [EQ-5D-5L]) in the two arms.

VII. To correlate baseline volume of disease on prostate-specific membrane antigen-positron emission tomography/computed tomography (PSMA-PET/CT) with baseline volume of disease on conventional imaging (CI).

VIII. To determine if baseline PSMA-PET/CT and CI are individually and jointly associated with OS, progression-free survival (PFS), PSA90 response, and PSA < 0.2 ng/ml after 6 months, and to estimate its clinical relevance when compared to these well characterized prognostic endpoints.

IX. To correlate 6-month PSA level with the presence/absence and volume of residual disease on PSMA-PET/CT after 6 months of doublet or triplet therapy.

X. To correlate the concordance of radiographic progression on CI versus PSMA-PET/CT at the time of PSA progression.

XI. To determine rPFS, time to castration resistance, OS based on thresholds of volume of disease, and prostate-specific membrane antigen (PSMA) uptake (standardized uptake value [SUV]) based on baseline PSMA-PET/CT scan.

XII. To compare rPFS, time to castration resistance, and OS between arms in patients with de novo metastatic disease having received primary directed radiation therapy.

XIII. To determine rPFS, time to castration resistance, and OS correlation with PSA response at 6 weeks and 6 months.

XIV. To compare the impact of treatment on aging trajectory, as measured by the change in Deficit-Accumulation Frailty Index (DAFI) from baseline, 6- and 12-months, in the two arms.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive ADT at the discretion of the investigator and apalutamide orally (PO) once daily (QD). Cycles repeat every 12 weeks in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo computed tomography (CT) scan or magnetic resonance imaging (MRI) and bone scan throughout the study. Patients may optionally undergo prostate-specific membrane antigen-positron emission tomography (PSMA-PET) scans and blood sample collection throughout the study.

ARM 2: Patients receive ADT at the discretion of the investigator and apalutamide PO QD. Cycles repeat every 12 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive docetaxel intravenously (IV) over 1 hour every 21 days for up to 6 doses. Additionally, patients undergo CT scan or MRI and bone scan throughout the study. Patients may optionally undergo PSMA-PET scans and blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 6 months for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of disease:

  * Histologically or cytologically confirmed adenocarcinoma of the prostate without small cell histology
* Must have had evidence of metastatic disease (American Joint Committee on Cancer [AJCC] metastasis [M]1 disease) based on conventional CT/MRI and/or bone scan. This will be defined as:

  * Bone metastases detected by CT, radionuclide technetium-99 (99Tc)- methylene bisphosphonate bone scan, or MRI as defined by PCWG3 criteria; OR
  * Non-pelvic lymph node metastases (measurable lymph nodes above the aortic bifurcation; lymph nodes are measurable if the short axis diameter is ≥ 15 mm) detected on CT or MRI as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Subjects with regional lymph node metastases only (nodes [N]1, below the aortic bifurcation) will not be eligible for the study; OR
  * Visceral or soft tissue metastases detected on CT or MRI as defined by RECIST version 1.1. Soft tissue/visceral lesions are measurable if the long axis diameter is ≥ 10 mm
  * Evidence of metastatic disease by PSMA-PET only and not visible by CT, radionuclide bone scan, or MRI will not satisfy eligibility criteria
* No metachronous low-volume disease (defined as recurrent metastatic disease after definitive treatment of prostate primary) and with ≤ 4 bone metastasis and no visceral metastasis on conventional imaging by CT, radionuclide 99Tc-biphosphonate bone scan, or MRI)
* Next generation sequencing (NGS) results from any tissue based Clinical Laboratory Improvement Act (CLIA) test must be available at the time of registration. NGS from soft tissue or visceral lesion if available is preferred. NGS from bone or primary prostate will be accepted. Patients with failed NGS testing are not eligible
* Prior treatment

  * ADT (luteinizing hormone-releasing hormone [LHRH] agonist/antagonist or orchiectomy) with or without first generation anti-androgen, or second-generation androgen receptor signaling inhibitor (ARSI) within 120 days of registration is permitted. No washout period will be needed for the first generation- androgen or ARSI prior to registration. Anti-androgen treatment is only permitted if used within 120 days of registration
  * No prior chemotherapy for prostate cancer
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ 1 x upper limit of normal (ULN) (Note: In subjects with Gilbert's syndrome, if total bilirubin is > 1.5 × ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤ 1 × ULN, subject may be eligible)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate transaminase [SGT]) ≤ 1.5 x upper limit of normal (ULN)
* Calculated (Calc.) creatinine clearance > 30 mL/min
* Serum potassium ≥ 3.5 mmol/L
* Comorbid conditions

  * Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
  * Leptomeningeal metastases: Patients with treated leptomeningeal metastases are eligible if follow-up brain imaging 30 days after central nervous system (CNS)-directed therapy shows no evidence of progression
  * HIV: Patients with known HIV infection on effective anti-retroviral therapy with undetectable viral load within 6 months prior to registration are eligible for this trial
  * Hepatitis B: For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
  * Hepatitis C: Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
  * No seizure or known condition that may pre-dispose to seizure (e.g. prior stroke within 1 year to randomization, brain arteriovenous malformation or condition requiring CNS surgery or radiation therapy)
  * Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association functional classification. To be eligible for this trial, patients should be class II or better. Any condition that in the opinion of the investigator, would preclude participation in this study. Patients with stable asymptomatic deep venous thromboembolism on stable anti-coagulation will be eligible
  * Hypertension: Subjects with uncontrolled hypertension as indicated by a resting systolic blood pressure (BP) >= 160 mmHg or diastolic BP >= 100 mmHg despite medical management are not permitted to register
  * Allergies: Subjects with known hypersensitivity to any of the study drugs, or excipients in the formulation of the study drugs are not permitted to register
* Concomitant medications

  * Chronic concomitant treatment with strong inhibitors of cytochrome P450 3A4 (CYP3A4) is not allowed on this study. Patients on strong CYP3A4 inhibitors must discontinue the drug prior to registration on the study. See Section 8.1.9 for more information
  * Chronic concomitant treatment with strong CYP3A4 inducers is not allowed. Patients must discontinue the drug 14 days prior to the start of study treatment
  * Medications known to lower the seizure threshold must be discontinued or substituted prior to study entry. See Section 8.1.9 for more information
* Patient agrees to use a condom (even men with vasectomies) and another effective method of birth control if having sex with a woman of childbearing potential or agrees to use a condom if having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug. Must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1260 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2031-11-11 (Estimated); Study Completion 2039-05-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From randomization to death due to any cause, assessed up to 10 years
  Will determine OS. To assess the potential OS benefit from the triplet therapy, a group sequential efficacy/futility monitoring design will be employed. The planned analyses for OS will be tested using a one-sided type 1 error rate of 0.025. An intent-to-treat approach will be used to evaluate OS between treatments. The stratified logrank test will be the primary analysis to compare OS between treatments. The Kaplan-Meier estimate will be used to evaluate the within treatment OS distributions. In addition, the proportional hazards model will be applied to assess the treatment comparison adjusting for important covariates in predicting OS.

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization to death due to any cause, assessed up to 10 years
  Will determine if the addition of docetaxel to androgen deprivation therapy and apalutamide improves OS for men whose cancers have alterations of P53, PTEN, or RB1. To assess the potential OS benefit from the triplet therapy, a group sequential efficacy/futility monitoring design will be employed. The planned analyses for OS will be tested using a one-sided type 1 error rate of 0.025. An intent-to-treat approach will be used to evaluate OS between treatments. The stratified logrank test will be the primary analysis to compare OS between treatments. The Kaplan-Meier estimate will be used to evaluate the within treatment OS distributions. In addition, the proportional hazards model will be applied to assess the treatment comparison adjusting for important covariates in predicting OS.
Radiographic progression | From randomization to first documentation of radiographic progressive disease or death due to any cause, assessed up to 10 years
  Will determine the time to radiographic progression- per Prostate Cancer Working Group (PCWG3) guidelines. Tumor response will be assessed utilizing imaging measurements, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. In this study, RECIST has been modified based on PCWG3 criteria, which are specific for this patient population.
Castration-resistant prostate cancer (CRPC) | Time to prostate-specific antigen progression with serum testosterone being at castrate level < 0.50 ng/mL, or the time to progression by soft tissue/visceral lesions or time to progression by bone lesions per PCWG3 guidelines, assessed up to 10 years
  Will determine the time to CRPC
Symptomatic skeletal event free survival (SSE-FS) | From randomization to first occurrence of SSE or death from any cause, assessed up to 10 years
  Will determine SSE-FS. An SSE is defined as external beam radiation therapy to relieve skeletal symptoms, or new symptomatic pathologic bone fracture, or occurrence of spinal cord compression or tumor-related orthopedic surgical intervention, whichever comes first
Worsening of physical symptoms of disease | up to 10 years
  Will determine the time to worsening of physical symptoms of disease based on functional assessment of cancer therapy / National Comprehensive Cancer Network prostate cancer symptom index 17 item questionnaire.
Incidence of adverse events | up to 10 years
  Will determine the safety and tolerability of the triplet versus doublet using Common Terminology Criteria for Adverse Events version 5.0.
Radiographic progression free survival (rPFS) | From randomization to first documentation of radiographic progressive disease or death due to any cause, assessed up to 10 years
  Will determine rPFS in patients by the stratification factors a) timing/volume of disease 1) metachronous high volume, 2) synchronous high volume and 3) synchronous low volume metastases on conventional imaging. Tumor response will be assessed utilizing imaging measurements, as defined by RECIST 1.1. In this study, RECIST has been modified based on PCWG3 criteria, which are specific for this patient population. Evaluation of rPFS will be assessed by the investigator.
OS | Will determine OS in patients by the stratification factors a) timing/volume of disease 1) metachronous high volume, 2) synchronous high volume and 3) synchronous low volume metastases on conventional imaging. To assess the potential OS benefit from the
  Will determine OS in patients by the stratification factors a) timing/volume of disease 1) metachronous high volume, 2) synchronous high volume and 3) synchronous low volume metastases on conventional imaging. To assess the potential OS benefit from the triplet therapy, a group sequential efficacy/futility monitoring design will be employed. The planned analyses for OS will be tested using a one-sided type 1 error rate of 0.025. An intent-to-treat approach will be used to evaluate OS between treatments. The stratified logrank test will be the primary analysis to compare OS between treatments. The Kaplan-Meier estimate will be used to evaluate the within treatment OS distributions. In addition, the proportional hazards model will be applied to assess the treatment comparison adjusting for important covariates in predicting OS.
Prostate specific antigen (PSA) 90 response rate | At 6 weeks and 6 months
  Will determine PSA 90 response rate.
Time to PSA progression | From randomization to the date of PSA progression based on PCWG3 criteria, assessed up to 10 years
  Will determine PSA progression. PSA progression is defined as a ≥ 25% increase above the nadir (lowest screening or baseline) value, which is confirmed by a second value 3 or more weeks later, and an increase in absolute value of ≥ 2 ng/mL above nadir, at least 12 weeks from baseline. Subjects without PSA progression as of database cut-off, whether or not surviving, will be censored at the last total PSA lab assessment date.
Objective response rate (ORR) | up to 10 years
  Will determine ORR in patients with measurable disease. Tumor response will be assessed utilizing imaging measurements, as defined by RECIST 1.1. In this study, RECIST has been modified based on PCWG3 criteria, which are specific for this patient population

OTHER OUTCOMES:
Estimates of treatment effect | up to 10 years.
  Estimates of treatment effect and the corresponding 95% confidence intervals (CIs) will be provided as follows (with an understanding that sometimes the CI or estimate will not be computable because of scant data):
  * Estimates of the OS hazard ratio and the corresponding 95% CIs by race.
  * Estimates of the OS hazard ratio and the corresponding 95% CIs by ethnicity.

CONTACTS AND LOCATIONS:
Locations (125):
- United States (125):
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente- Modesto MOB II, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Bayhealth Hospital Sussex Campus, Milford, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Community Medical Center, Missoula, Montana
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Jefferson Cherry Hill Hospital, Cherry Hill, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Froedtert and MCW Moorland Reserve Health Center, New Berlin, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided